CLINICAL TRIAL: NCT03536247
Title: Prospective Randomized Trial of Cholangioscopy Guided Intraductal Lithotripsy Versus Papillary Balloon Dilation for the Endoscopic Treatment of Large Bile Duct Stones
Brief Title: Papillary Balloon Dilation Versus Intraductal Lithotripsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Ara Sahakian, Assistant Professor of Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-17-00448
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Choledocholithiasis
Keywords: bile duct stones; choledocholithiasis; ERCP; endoscopic retrograde cholangiopancreatograhy
MeSH Terms: conditions — Choledocholithiasis; Cholecystolithiasis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized using a pre-generated randomization schedule with concealed allocation in a 1:1 assignment to initial cholangioscopy guided lithotrispy or papillary dilation. Randomization will be blocked in groups of 12.
Who Masked: Participant
Masking Description: Participants in the study will be blinded to treatment arm. Care providers and Investigators will be unblinded to treated arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraductal lithotripsy (Active Comparator): Cholangioscopy enables therapeutic intervention including intracorporeal electro-hydraulic and laser lithotripsy for biliary stone disease with favorable efficacy and safety.
  Interventions: Procedure: Initial therapy with intraductal lithotripsy
- Papillary Balloon dilation (Active Comparator): Balloon dilation of the Ampulla of Vater after a small sphincterotomy is an alternative technique that allows for removal of large bile duct stones in a safe and effective manner.
  Interventions: Procedure: Initial therapy with papillary balloon dilation

INTERVENTIONS:
Procedure: Initial therapy with papillary balloon dilation — patients will first undergo papillary dilation
  Other Names: papillary dilation
  Arms: Papillary Balloon dilation
Procedure: Initial therapy with intraductal lithotripsy — patients will first undergo intraductal laser or electrohydraulic lithrotripsy
  Arms: Intraductal lithotripsy

SUMMARY:
Our aim is to compare the efficacy, safety, procedural time required, and costs of a strategy initially employing cholangioscopy guided intraductal lithotripsy (laser/electrohydraulic lithtripsy (EHL)) versus a strategy initially using papillary dilation for removal of large bile duct stones.

DETAILED DESCRIPTION:
The study will be a prospective single blind randomized comparative trial. All patients presenting with choledocholithiasis will be considered for the study. If their ultrasound, computed tomography, or magnetic resonance imaging demonstrates a large stone (>1cm) and they do not fulfill the exclusion criterion they will be eligible for the study. If a prior Endoscopic retrograde cholangiopancreatography (ERCP) demonstrates a stone >1cm, which could not be removed with standard methods, they will also be eligible. Randomization will be stratified based on whether or not the procedure is a first or repeat ERCP

Patients will be randomized using a computer generated randomization schedule with concealed allocation in a 1:1 assignment (allocation ratio) to initial cholangioscopy guided lithoripsy versus initial papillary dilation. Randomization will be blocked in groups of 12.

In those randomized to cholangioscopy-guided lithotripsy, the procedure will be performed in the standard manner using a single operator cholangioscopy system and a holmium laser or EHL (dependent on availability). Those in the papillary dilation arm will undergo the standard approach using the combined papillary dilation balloon sphincterotomy system. The patients will be blinded as to treatment arm.

"Conventional" methods including mechanical lithotripsy or stent placement may be used to remove stones/debris in combination with the specified intervention, as is done for standard clinical care. Use of these strategies will be recorded

If stone removal fails with the assigned strategy, this will be considered failure of the assigned intervention. This decision will be made by the attending endoscopist and recorded. The patient will then crossover into the other treatment arm.

The primary outcome will be complete stone clearance in the first study procedure by the assigned method. Additional outcomes will be total procedure time, cost of equipment, and number and type of complications. Additional ERCP may be needed for complete removal in some cases (i.e. complete removal in first attempt is not possible), thus we will also compare the number of ERCP needed for final stone clearance and whether stone removal is eventually achieved by endoscopic methods (comparison will be on an intention to treat basis). Additionally, if patients require surgical stone removal for the standard clinical indication in the case that endoscopic strategies are not successful, this will be recorded.

The patients will be followed clinically by the principal investigator assisted by a research coordinator on days 1,7 and 30 post procedures. This will be done as a brief follow up visit if the patient is still hospitalized or by telephone call thereafter.

Thus, all procedures performed in this study represent standard clinical care, which would be used even if the patients did not take part in the study, except that the initial choice to use cholangioscopy guided lithotripsy versus papillary dilation will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Undergoing ERCP at LAC+Medical Center or Keck Hospital of USC for the standard indication of bile duct stones with evidence of a large stone (>1cm) demonstrated either on Ultrasound, computed tomography, prior ERCP, or magnetic resonance imaging.

Exclusion Criteria:

* Patients Under the age of 18
* Patients with biliary malignancy
* Prior biliary diversion surgery
* Prior gastric bypass surgery
* Patients who are incarcerated
* Patients who are unable to give consent
* Patients who pregnant

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
First procedure stone clearance | 2 hours
  Entire stone[s] removed in first procedure

SECONDARY OUTCOMES:
Adverse Events | 1 week
  Pancreatitis, bleeding, perforation, infection
Procedure Time | 2 hours
  Length of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ara Sahakian, MD, Principal Investigator — University of Southern California; James Buxbaum, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles County + USC Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang WH, Chu CH, Wang TE, Chen MJ, Lin CC. Outcome of simple use of mechanical lithotripsy of difficult common bile duct stones. World J Gastroenterol. 2005 Jan 28;11(4):593-6. doi: 10.3748/wjg.v11.i4.593. PMID 15641153
- [Background] Moon JH, Ko BM, Choi HJ, Hong SJ, Cheon YK, Cho YD, Lee JS, Lee MS, Shim CS. Intraductal balloon-guided direct peroral cholangioscopy with an ultraslim upper endoscope (with videos). Gastrointest Endosc. 2009 Aug;70(2):297-302. doi: 10.1016/j.gie.2008.11.019. Epub 2009 Apr 25. PMID 19394010
- [Background] Lee JG. Diagnosis and management of acute cholangitis. Nat Rev Gastroenterol Hepatol. 2009 Sep;6(9):533-41. doi: 10.1038/nrgastro.2009.126. Epub 2009 Aug 4. PMID 19652653
- [Background] Kim HI, Moon JH, Choi HJ, Lee JC, Ahn HS, Song AR, Lee TH, Cho YD, Park SH, Kim SJ. Holmium laser lithotripsy under direct peroral cholangioscopy by using an ultra-slim upper endoscope for patients with retained bile duct stones (with video). Gastrointest Endosc. 2011 Nov;74(5):1127-32. doi: 10.1016/j.gie.2011.07.027. Epub 2011 Sep 29. PMID 21963070
- [Background] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903
- [Background] Stefanidis G, Viazis N, Pleskow D, Manolakopoulos S, Theocharis L, Christodoulou C, Kotsikoros N, Giannousis J, Sgouros S, Rodias M, Katsikani A, Chuttani R. Large balloon dilation vs. mechanical lithotripsy for the management of large bile duct stones: a prospective randomized study. Am J Gastroenterol. 2011 Feb;106(2):278-85. doi: 10.1038/ajg.2010.421. Epub 2010 Nov 2. PMID 21045816
- [Background] Itoi T, Itokawa F, Sofuni A, Kurihara T, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Moriyasu F. Endoscopic sphincterotomy combined with large balloon dilation can reduce the procedure time and fluoroscopy time for removal of large bile duct stones. Am J Gastroenterol. 2009 Mar;104(3):560-5. doi: 10.1038/ajg.2008.67. Epub 2009 Jan 27. PMID 19174779
- [Background] Itoi T, Sofuni A, Itokawa F, Kurihara T, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Umeda J, Moriyasu F. New large-diameter balloon-equipped sphincterotome for removal of large bile duct stones (with videos). Gastrointest Endosc. 2010 Oct;72(4):825-30. doi: 10.1016/j.gie.2010.06.018. PMID 20883862
- [Background] Kiriyama S, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Yokoe M, Kimura Y, Tsuyuguchi T, Itoi T, Yoshida M, Miura F, Yamashita Y, Okamoto K, Gabata T, Hata J, Higuchi R, Windsor JA, Bornman PC, Fan ST, Singh H, de Santibanes E, Gomi H, Kusachi S, Murata A, Chen XP, Jagannath P, Lee S, Padbury R, Chen MF, Dervenis C, Chan AC, Supe AN, Liau KH, Kim MH, Kim SW; Tokyo Guidelines Revision Committee. TG13 guidelines for diagnosis and severity grading of acute cholangitis (with videos). J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):24-34. doi: 10.1007/s00534-012-0561-3. PMID 23307001